CLINICAL TRIAL: NCT05128461
Title: The Effectiveness of Modified-Constraint Induced Movement Therapy Based Telerehabilitation in Stroke Patients
Brief Title: The Effectiveness of Telerehabilitation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fettah Saygılı, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-Stroke-CIMT-Telerehab.
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: Stroke; Telerehabilitation; modified-Constraint Induced Movement Therapy; Upper Extremity
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups as exercise group and control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The group will receive modified-Constraint Induced Movement Therapy via telerehabilitation and a home exercise program.
  Interventions: Other: Exercise; Other: Home program
- Control group (Active Comparator): The group only will be given a home exercise program.
  Interventions: Other: Home program

INTERVENTIONS:
Other: Exercise — M-CIMT-based telerehabilitation will be implemented.
  Arms: Exercise Group
Other: Home program — Lower and upper extremity exercises and gait training exercises selected according to the Bobath approach will be given as a home program consisting of 10 same exercises.

SUMMARY:
Stroke, according to the definition of the World Health Organization (WHO); It is a syndrome characterized by a rapid settlement of signs and symptoms of focal loss of cerebral function without a cause other than vascular causes. As it is known, it is important for patients to regain functional skills in the upper extremities after stroke. Modified-Constraint Induced Movement Therapy (m-CIMT) is a versatile neurorehabilitation technique that aims to improve motor function in the hemiparetic upper extremity and increase its use in daily life activities. However, as in the Covid-19 pandemic, patients cannot always reach rehabilitation services. In such cases, telerehabilitation is a treatment option. There are a limited number of studies in which m-CIMT is applied according to the principle of telerehabilitation, which has become a necessity, especially due to the Covid-19 pandemic. Therefore, the aim of this study is to examine the effects of m-CIMT on upper extremity motor functions in stroke patients.

DETAILED DESCRIPTION:
This study is a randomized controlled study. The patients will be randomly divided into two groups as exercise and control. Patients in both groups will be given lower-upper extremity exercises and gait training exercises selected according to the Bobath approach as a home program consisting of 10 exercises to be applied 5 days a week for 3 weeks. All patients will perform the same exercises. In addition, the exercise group will receive Modified-Constraint Induced Movement Therapy (m-CIMT) based telerehabilitation via video conferencing 5 days a week for 3 weeks. Patients in the m-CIMT group will be asked to restrict the movements of their less affected hands by using mitt for 5 hours a day/ 5 days a week for 3 weeks while the patients are awake. Evaluations for both groups will be made by a physiotherapist blinded to the study twice, at the beginning and 3 weeks later. As outcome measures functional performance, hand strength, activities of daily living and quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Being diagnosed with stroke for the first time by a doctor
* Having been diagnosed with stroke at least 1 month ago
* Mini-Mental Test Score more than or equal 24
* In the upper extremities; Starting from the angle of full flexion, wrist extension of at least 20° or more, thumb extension or abduction of at least 10°, minimum extension of all other fingers at the metacarpophalangeal and interphalangeal joints
* Having less than 2.5 points in the pre-treatment evaluation from both parts of MAG-28
* Being able to stand for 2 minutes without any help by using the upper extremity as a support tool when necessary.
* Absence of severe pain to affect the treatment
* Absence of severe spasticity to affect the treatment (spasticity in any joint of the upper extremity ≤ 2 according to the Modified Ashworth Scale)

Exclusion Criteria:

* Any orthopedic, vision, hearing or perception problems that may affect the research results
* Having an additional neurological, cardiovascular, pulmonary or hormonal disorder that would prevent participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Upper extremity motor ability-Baseline | Assessment will be conducted before the intervention.
  Wolf Motor Function Test
Upper extremity motor ability-Post intervention | Assessment will be conducted immediately after the intervention.
  Wolf Motor Function Test
Upper extremity motor function-Baseline | Assessment will be conducted before the intervention.
  The Fugl-Meyer Assessment of the Upper Extremity
Upper extremity motor function-Post intervention | Assessment will be conducted immediately after the intervention.
  The Fugl-Meyer Assessment of the Upper Extremity
Activities of daily living related to the upper extremity-Baseline | Assessment will be conducted before the intervention.
  Motor Activity Log-28 (MAL-28) The minimum score that can be obtained from this scale is 0, and the maximum score is 5. Higher scores mean that the level of use and quality of use is better.
Activities of daily living related to the upper extremity-Post intervention | Assessment will be conducted immediately after the intervention.
  Motor Activity Log-28 (MAL-28) The minimum score that can be obtained from this scale is 0, and the maximum score is 5. Higher scores mean that the level of use and quality of use is better.
Voluntary movement and mobility-Baseline | Assessment will be conducted before the intervention.
  Stroke Rehabilitation Assessment of Movement (STREAM)
Voluntary movement and mobility-Post intervention | Assessment will be conducted immediately after the intervention.
  Stroke Rehabilitation Assessment of Movement (STREAM)

SECONDARY OUTCOMES:
Isometric hand strength-Baseline | Assessment will be conducted before the intervention.
  J-Tech™
Isometric hand strength-Post intervention | Assessment will be conducted immediately after the intervention.
  J-Tech™
Isometric pinch strength-Baseline | Assessment will be conducted before the intervention.
  Baseline® pinch meter
Isometric pinch strength-Post intervention | Assessment will be conducted immediately after the intervention.
  Baseline® pinch meter
manual dexterity performance-Baseline | Assessment will be conducted before the intervention.
  nine-hole peg test (9-HTP)
manual dexterity performance-Post intervention | Assessment will be conducted immediately after the intervention.
  nine-hole peg test (9-HTP)
level of independence in activities of daily living-Baseline | Assessment will be conducted before the intervention.
  Functional Independence Measure
level of independence in activities of daily living-Post intervention | Assessment will be conducted immediately after the intervention.
  Functional Independence Measure

CONTACTS AND LOCATIONS:
Overall Officials: Fettah SAYGILI, PT, M.Sc., Study Chair — Research Assistant; Arzu Güçlü-Gündüz, PT, PhD., Study Director — Professor
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD data but when the statistical analysis of all data is made, all results will be shared.

REFERENCES:
- See also: Related info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7502810/